CLINICAL TRIAL: NCT03225898
Title: Upper- and Lower-body Resistance Exercise With and Without Blood Flow Restriction on Hemodynamics and Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, J. Derek Kingsley, Assistant Professor, Kent State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-285
Record Dates: First submitted 2017-07-10; First posted 2017-07-21 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Endothelial Dysfunction; Autonomic Dysfunction
Keywords: blood flow restriction; resistance exercise
MeSH Terms: conditions — Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise with Blood flow restriction (Experimental): Subjects will perform 4 sets with 30, 15, 15, 15 repetitions at 30% 1RM.
  Interventions: Other: Resistance Exercise with Blood Flow Restriction
- High-intensity resistance exercise (Active Comparator): Subjects will perform 4 sets of 8 repetitions at 70% 1RM.
  Interventions: Other: High-intensity Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise with Blood Flow Restriction — A cuff will be used to restrict blood flow to the extremities.
  Other Names: KATTSU
  Arms: Resistance Exercise with Blood flow restriction
Other: High-intensity Resistance Exercise — Participants will follow a conventional resistance exercise regime.
  Arms: High-intensity resistance exercise

SUMMARY:
The American College of Sports Medicine (ACSM) recommends that resistance exercise performed at greater than 70% one repetition maximum (1 RM) is necessary to induce strength gains and muscular hypertrophy (ACSM, 2009). However, previous work has shown resistance exercise at high intensity increases the rate of injury. Blood flow restriction (BFR) exercise is a method that is used to compress the blood vessels to the exercising muscle in order to reduce blood flow to the limb with the use of low-intensity resistance. Researchers have suggested that resistance exercise at intensities as low as 20-30% 1-repetition maximum with BFR increases in muscle mass, muscular endurance, and gains in strength. However, the acute heart and blood vessel changes in response to BFR are not clear. Work by our laboratory (Tai et al., 2016) has demonstrated that immediately following acute resistance exercise at moderate intensity (75% 1 RM) without BFR, there are no changes in aortic and brachial systolic and diastolic blood pressure (BP), but there are increases in the pressure of the reflective wave (augmentation pressure). This suggests that the arterial wall is stiff, and may in turn result in thickening of the arterial wall. However, the data are limited and these responses may not be universally accepted. In addition, these studies used primarily lower-body resistance exercises (squat, leg extension, and leg flexion), and did not assess changes in heart and blood vessel function. Previous researchers have demonstrated that upper-body exercise induces higher BP and heart rate (HR) than lower-body exercise. However, the effects of upper- and lower-body resistance exercise with BFR on heart and blood vessel function are still unclear. Therefore, understanding the effects of upper- and lower-body resistance exercise with BFR on heart and blood vessel function using weight machines, specifically the chess press, latissimus dorsi pulldown, knee extension, and knee flexion may significant impact how the resistance training program is prescribed.

DETAILED DESCRIPTION:
Participants will come to the Cardiovascular Dynamics Laboratory at Kent State University for 4 separate visits. On the first visit, participants will undergo an orientation and decide if they want to sign the informed consent. If they decide to consent, they will be assigned randomly to either upper- or lower-body group, and fill out Physical Activity Readiness Questionnaire (PAR-Q) and Health Participant Questionnaire then be measured for height, weight, body composition (7-sites skin fold), arterial occlusion pressure (determine the pressure that occlude blood flow using a doppler device on brachial or femoral artery, and a 13-cm nylon cuff at the proximal end of right arm or right leg then inflate the cuff to 50 mmHg and increases by 1 mmHg per second until the doppler device cannot detect blood flow) and 1 RM which they will move maximum amount of weight 1 time through a full range of motion on the chess press and latissimus dorsi pulldown or knee extension and knee flexion. A certified strength and conditioning specialist will adjust the form, spot the lifts, and provide feedback if needed. The second visit consists of 1-repetition maximum verification that participants will be measured 1-repetition maximum on the chess press and latissimus dorsi pulldown or knee extension and knee flexion again to ensure their maximal strength. For the third and fourth visits, the participants will come to the Cardiovascular Dynamics Laboratory to have their responses to either acute upper- or lower-body resistance exercise with and without BFR quantified. Participants will arrive at the laboratory having avoided caffeine, alcohol, and strenuous exercise for 24 hours, and at least 3 hours without food before data collection. Participants will have their hemodynamics and vascular function measured before and after either acute upper- or lower-body resistance exercise with or without BFR. Hemodynamic measurements will include pulse wave analysis (PWA) using a SphygmoCor (AtCor Medical, Sydney, Australia) device. Heart rate and blood pressure will be monitored using 3 leads electrocardiograph (ECG) and on the middle finger of the right hand, respectively. A 5-minute ECG will be collected, and participants will be breathing with a metronome at the rate of 12 breaths/minute. PWA provides information about aortic and brachial systolic and diastolic BP, as well as measures of wave reflection that give insight into central arterial modulation such as augmentation pressure and the augmentation index. BP will be measured twice separated by 1 minute by an oscillometric device. After that the investigators will assess vascular function via pulse wave velocity. During PWA measurements, there will be cuffs on right arm and right leg, and a tonometer will be placed on the carotid artery on the neck. Peripheral arterial mechanics will be measured by strain gauge plethysmography (EC-6; DE Hokanson Inc., Bellevue, WA, USA) on the forearm close to the elbow in order to determine forearm blood flow and vasodilatory capacity (peak blood flow). There will be cuffs on the upper left arm and on the left wrist. The wrist Cuff will be inflated to 220 mmHg 1 minute prior to data collection and throughout. The Upper arm cuff will be inflated to 50 mmHg to occlude venous flow for measurement of arterial flow. Ninety seconds of measurement of flow will occur. Once this is completed, the cuff on the upper arm will be inflated to 220 mmHg for 5 minutes to occlude blood flow. After that, the pressure in the cuff will be released and measurements of blood flow will be taken for the next 3 minutes with the wrist cuff will be inflated to 220 mmHg 1 minute prior to data collection and throughout. The upper-(chess press and latissimus dorsi pulldown) and lower-body (knee extension and knee flexion) resistance exercise with BFR will consists of 4 sets of 30, 15, 15, and 15 repetitions at 30% 1 RM with 30 seconds rest between sets and 2 minutes rest between exercises. The upper- and lower-body resistance exercise without BFR will consists of 4 sets of 8 repetitions at 70% 1 RM with 60 seconds rest between sets and 2 minutes rest between exercises. Participants' arms or legs will be wrapped using elastic cuffs at the most proximal limbs. At 40% of arterial occlusion pressure will be used to induce BFR. Three minutes warm up and three minutes cool down on the cycle ergometer will be given before and after resistance exercise. Immediately after completion of the acute bouts of resistance exercise, the investigators will assess PWA and ECG at 10, 20, 30, 40, 50, and 60 minutes post exercise, and BF at 20 and 60 minutes post exercise.

ELIGIBILITY:
Inclusion Criteria:

* 3 days per week of resistance training for 1 year
* 18-30 years of age

Exclusion Criteria:

* include a recent smoking history (< 6 months)
* obesity (defined as a body mass index ≥ 30 kg/m2)
* skeletal and orthopedic injuries
* cancer
* known cardiovascular disease
* open wounds
* history of blood clots
* metabolic disease
* uncontrolled hypertension (resting brachial BP ≥ 140/90 mmHg)
* pregnancy, planning to get pregnant
* taking any medications or supplements known to affect blood pressure, heart rate, or vascular function

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-06-13 (Estimated); Study Completion 2018-06-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Autonomic Modulation over 1 hour | Rest, 10 min, 20 min, 30 min, 40 min, 50 min, 60 min post exercise
  Heart rate variability

SECONDARY OUTCOMES:
Change from Baseline Endothelial Function over 1 hour | Rest, 10 min, 20 min, 30 min, 40 min, 50 min, 60 min post exercise
  Pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: J. Derek Kingsley, PhD, Principal Investigator — Kent State University
Locations (1):
- Cardiovascular Dynamics Laboratory, Kent, Ohio, United States

REFERENCES:
- [Background] Madarame H, Neya M, Ochi E, Nakazato K, Sato Y, Ishii N. Cross-transfer effects of resistance training with blood flow restriction. Med Sci Sports Exerc. 2008 Feb;40(2):258-63. doi: 10.1249/mss.0b013e31815c6d7e. PMID 18202577
- [Background] Takarada Y, Sato Y, Ishii N. Effects of resistance exercise combined with vascular occlusion on muscle function in athletes. Eur J Appl Physiol. 2002 Feb;86(4):308-14. doi: 10.1007/s00421-001-0561-5. PMID 11990743
- [Background] Rossow LM, Fahs CA, Sherk VD, Seo DI, Bemben DA, Bemben MG. The effect of acute blood-flow-restricted resistance exercise on postexercise blood pressure. Clin Physiol Funct Imaging. 2011 Nov;31(6):429-34. doi: 10.1111/j.1475-097X.2011.01038.x. Epub 2011 Jul 7. PMID 21981453
- [Background] Figueroa A, Vicil F. Post-exercise aortic hemodynamic responses to low-intensity resistance exercise with and without vascular occlusion. Scand J Med Sci Sports. 2011 Jun;21(3):431-6. doi: 10.1111/j.1600-0838.2009.01061.x. Epub 2010 Jan 31. PMID 20136757

DOCUMENTS (1):
  • Informed Consent Form (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03225898/ICF_000.pdf